CLINICAL TRIAL: NCT01207609
Title: A Prospective Study to Evaluate the Safety and Efficacy of the Laparoscopic Gastric Plication Operation for Patients With Severe or Morbid Obesity
Brief Title: Laparoscopic Gastric Plication Operation for Patients With Severe or Morbid Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ponce, Jaime, M.D. (Individual)
Responsible Party: Principal Investigator, Jaime Ponce MD, Director for Bariatric Surgery, Ponce, Jaime, M.D.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-9-001
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Morbid Obesity
Keywords: Obesity; Morbid Obesity; Bariatric Surgery; Laparoscopic Gastric Plication
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laparoscopic Gastric Plication (Experimental): Collect data prospectively on the safety and efficacy of the Laparoscopic Gastric Plication operation for 50 patients with Severe or Morbid Obesity
  Interventions: Procedure: Laparoscopic Gastric Plication

INTERVENTIONS:
Procedure: Laparoscopic Gastric Plication — The procedure is performed laparoscopic. The greater curvature of the stomach is separated from the greater omentum using a harmonic scalpel starting approximately 3-5 cm from the pylorus and ending at the angle of His. As needed, adhesions to the posterior surface of the stomach may be transected. At least two rows stitches will be placed laparoscopically about the greater curvature of the stomach starting at or near the angle of His and ending in the antrum. A calibration tube or endoscope will be used to maintain a lumen during the procedure, ensuring one exists after the procedure.
  Other Names: Laparoscopic Greater Curvature Plication; Vertical Gastric Plication; Gastric Sleeve Plication

SUMMARY:
The purpose of this study is to collect data prospectively on the safety and efficacy of the Laparoscopic Gastric Plication operation for patients with Severe or Morbid Obesity.

The 95% confidence interval for average percentage of weight loss and body mass index will be computed at 6 months, one year and then annually. Analysis of comorbid conditions changes, quality of life and adverse events will be performed. With 50 subjects in the study, limited power is expected and no formal hypothesis testing will be performed.

DETAILED DESCRIPTION:
The laparoscopic gastric plication (LGP) is a new restrictive bariatric surgical technique that has the potential to eliminate the complications associated with other restrictive procedures (i.e., gastric banding, sleeve gastrectomy) by creating a restriction without the use of an implant and without performing gastric resection. LGP is notably similar to a sleeve gastrectomy in that it generates a gastric tube by means of eliminating the greater curvature but does so without gastric resection.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 60 years
* BMI 35-39.9 kg/m2 with one or more severe co-morbid conditions or BMI 40-55 kg/m2
* Willingness to comply with dietary restrictions required by the protocol
* History of obesity for at least 5 years
* History of at least 6 months of documented failures with traditional non-surgical weight loss methods
* Willingness to follow protocol requirements which include: signing the informed consent form, completing routine follow-up visits for the study duration, and completing all pre- and post-operative laboratory and diagnostics tests in addition to the quality of life questionnaire
* If female with childbearing potential, using an appropriate form of contraception

Exclusion Criteria:

* Age less than 18, age greater than 60
* Pregnancy
* History of major depressive disorder or psychosis
* Previous bariatric surgery or previous gastric surgery
* Presence of achalasia
* Any condition that, in the judgment of the investigator, would place a subject at undue risk, or could potentially compromise the results or interpretation of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2010-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Percent of excess weight loss | 3 years
  The primary efficacy variable is weight loss, which is measured in pounds and evaluated in terms of % excess weight loss (EWL) and body mass index (BMI), both of which will be measured at each follow-up visit.
  Percent EWL is calculated by the following equation: [Weight Lost]/ [(Pre-op Weight)-(Ideal Body Weight)]. BMI is calculated by the equation: Weight (kg) divided by Height (m) squared [kg/m2].

SECONDARY OUTCOMES:
Status of comorbid conditions | 3 years
  Improvement, resolution or worsening of pre-operative co-morbidities will be evaluated and reported at one year and annually up to 3 years. Status will be evaluated according to the necessity of medications to maintain normal physiologic values such as fasting serum glucose in diabetic patients, normal blood pressure in hypertensive patients, and use of a CPAP machine for patients with obstructive sleep apnea.
Changes in quality of life scores from base line | 3 years
  Status of quality of life will be evaluated objectively with a standardized SF-36 Health Survey
Adverse events | 3 years
  Adverse events are intended to be volunteered by subjects or observed by the investigator. All adverse events are to be recorded on appropriate case report forms.

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ponce, MD, Principal Investigator — Hamilton Medical Center
Locations (2):
- United States (2):
  - Hamilton Medical Center, Dalton, Georgia
  - Chattanooga Bariatrics, Chattanooga, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramos A, Galvao Neto M, Galvao M, Evangelista LF, Campos JM, Ferraz A. Laparoscopic greater curvature plication: initial results of an alternative restrictive bariatric procedure. Obes Surg. 2010 Jul;20(7):913-8. doi: 10.1007/s11695-010-0132-0. PMID 20407932